CLINICAL TRIAL: NCT04653935
Title: Fully-remote Trial of a Self-management App for Those Living With Sjögren's Syndrome: Randomised Pilot and Feasibility Study
Brief Title: Pilot Feasibility Study of a Sjögren's Syndrome Self-management App
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northumbria University (Other)
Collaborators: Newcastle University (Other); Teesside University (Other); Versus Arthritis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 118742
Record Dates: First submitted 2020-11-24; First posted 2020-12-04 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-11

CONDITIONS: Sjogren's Syndrome
Keywords: Self-management; Smartphone; Autoimmune; Rheumatology
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full app with all app components (Experimental): Users receive app that contains all intervention components including: Symptom and Lifestyle information, Energy management, Goal Setting, Managing Difficult Times, Assertiveness and Communication Skills.
  Interventions: Behavioral: Self-management app with all intervention components
- Control minimal app with information component only (Active Comparator): Users receive app that contains only Symptom and Lifestyle information, and cannot see other intervention components.
  Interventions: Behavioral: Self-management app with Information component only

INTERVENTIONS:
Behavioral: Self-management app with all intervention components — A behavioural self-management app, containing multiple cognitive- and behavioural self-management techniques for those living with Sjögren's syndrome. The intervention is comprised of several components and modules that holistically target several key symptoms: fatigue, sleep disturbances, chronic pain, and dryness. The app has been developed using user-centred methods, and is theory- and evidence-based.
  Other Names: Sjogo app
  Arms: Full app with all app components
Behavioral: Self-management app with Information component only — self-management app for those with Sjögren's syndrome, includes Symptom and Lifestyle Information, only.
  Other Names: Sjogo app_information only
  Arms: Control minimal app with information component only

SUMMARY:
This study investigates the feasibility of a fully remote effectiveness evaluation of a self-management smartphone application for those with Sjogren's syndrome.

DETAILED DESCRIPTION:
The aim of this study is to pilot and assess the feasibility of a fully remote effectiveness evaluation of a smartphone self-management app for those living with Sjogren's syndrome.

The fully-remote evaluation will involve minimal contact with researchers. Potential participants will be recruited internationally online through social media and mailing lists for Sjogren's syndrome support groups. Adverts will direct people to download the self-management app on app stores (Apple App Store and Google Play). The app has been designed to automate all study procedures, by guiding users through the following processes: screening, informed consent, randomisation, and the collection of outcome data through in-app surveys sent at 0, 5, and 10 weeks. Users will be randomised to receive the full intervention or a control:

* Intervention group: full version of the app containing multiple behavioural components: Symptom and Lifestyle Information, Energy Management, Goal Setting, Managing Difficult Times, Assertiveness and Communication Skills.
* Control Group: minimal version of the app containing only the Symptom and Lifestyle Information component.

To pilot and assess the feasibility of the planned methodology, and inform the design of a future definitive randomised control trial of the app, the primary objectives of this study are to: characterise users (i.e. international recruitment and consent rates), and test screening, randomisation and data collection procedures (i.e. outcome measure completion rates and score variability). The secondary objectives are to explore app engagement patterns (using log data) and the acceptability of the study procedures and the app (using remote semi-structured interviews).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosed with either Primary or Secondary Sjogren's syndrome (self-report)
* Own an iPhone or Android smartphone

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 996 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Number of people downloading the app | Through to completion of data collection period of up to 6 months
  Total number of people who download the app from App Stores
Percentage of eligible users (denominator is number downloading) | Through to completion of data collection period up to 6 months
  Proportion of users who have downloaded the app that are eligible to participate
Percentage of consenting users (denominator is number eligible) | Through to completion of data collection period up to 6 months
  Proportion of those who are eligible to participate that consented to take part in the study
Percentage of randomised users (denominator is number eligible) | Through to completion of data collection period up to 6 months
  Proportion of those who are eligible to participate that complete all surveys at week 0 and then automatically randomised to one of two app versions.
Percentage of retained users (denominator is number consenting) at 5 weeks | Through to completion of data collection period up to 6 months
  Proportion of those who those who consent to participate that complete all surveys at 5 weeks
Percentage of retained users (denominator is number consenting) at 10 weeks | Through to completion of data collection period up to 6 months
  Proportion of those who those who consent to participate that complete all surveys at 10 weeks
ICECAP-A Completion rate (denominator is number consenting) at 0 weeks | 0 weeks from date of consent
  Percentage of those who consent to take part that complete all 5 questions of ICECAP-A survey
ICECAP-A Completion rate (denominator is number consenting) at 5 weeks | 5 weeks from date of consent
  Percentage of those who consent to take part that complete all 5 questions of ICECAP-A survey
ICECAP-A Completion rate (denominator is number consenting) at 10 weeks | 10 weeks from date of consent
  Percentage of those who consent to take part that complete all 5 questions of ICECAP-A survey
ICECAP-A Mean Score at 0 weeks | 0 weeks from date of consent
  Average score on "ICECAP-A" Quality of Life Measure across participants
ICECAP-A Mean Score at 5 weeks | 5 weeks from date of consent
  Average score on "ICECAP-A" Quality of Life Measure across participants
ICECAP-A Mean Score at 10 weeks | 10 weeks from date of consent
  Average score on "ICECAP-A" Quality of Life measure across participants
ICECAP-A Standard Deviation of Mean Score at 0 weeks | 0 weeks from date of consent
  Standard deviation around Mean Score on "ICECAP-A" Quality of Life Measure across participants
ICECAP-A Standard Deviation of Mean Score at 5 weeks | 5 weeks from date of consent
  Standard deviation around Mean Score on "ICECAP-A" Quality of Life Measure across participants
ICECAP-A Standard Deviation of Mean Score at 10 weeks | 10 weeks from date of consent
  Standard deviation around Mean Score on "ICECAP-A" Quality of Life Measure across participants
ESSPRI Completion Rate (denominator is number consenting) at 0 weeks | 0 weeks from date of consent
  Percentage of those who consent to take part that complete all 3 questions of ESSPRI symptom severity survey (assessing dryness, fatigue and pain symptoms).
ESSPRI Completion Rate (denominator is number consenting) at 5 weeks | 5 weeks from date of consent
  Percentage of those who consent to take part that complete all 3 questions of ESSPRI survey (assessing dryness, fatigue and pain symptoms).
ESSPRI Completion Rate (denominator is number consenting) at 10 weeks | 10 weeks from date of consent
  Percentage of those who consent to take part that complete all 3 questions of ESSPRI symptom severity survey (assessing dryness, fatigue and pain symptoms).
ESSPRI Mean Score at 0 weeks | 0 weeks from date of consent
  Average score on "ESSPRI" symptom severity measure across participants
ESSPRI Mean Score at 5 weeks | 5 weeks from date of consent
  Average score on "ESSPRI" symptom severity measure across participants
ESSPRI Mean Score at 10 weeks | 10 weeks from date of consent
  Average score on "ESSPRI" symptom severity measure across participants
ESSPRI Standard Deviation of Mean Score at 0 weeks | 0 weeks from date of consent
  Standard deviation around Mean Score on ESSPRI symptom severity measure across participants
ESSPRI Standard Deviation of Mean Score at 5 weeks | 5 weeks from date of consent
  Standard deviation around Mean Score on ESSPRI symptom severity measure across participants
ESSPRI Standard Deviation of Mean Score at 10 weeks | 10 weeks from date of consent
  Standard deviation around Mean Score on ESSPRI symptom severity measure across participants
MFIS-5 Completion Rate (denominator is number consenting) at 0 weeks | 0 weeks from date of consent
  Percentage of those who consent to take part that complete all 5 questions of the Modified Fatigue Impact Scale
MFIS-5 Completion Rate (denominator is number consenting) at 5 weeks | 5 weeks from date of consent
  Percentage of those who consent to take part that complete all 5 questions of the Modified Fatigue Impact Scale
MFIS-5 Completion Rate (denominator is number consenting) at 10 weeks | 10 weeks from date of consent
  Percentage of those who consent to take part that complete all 5 questions of the Modified Fatigue Impact Scale
MFIS-5 Mean Score at 0 weeks | 0 weeks from date of consent
  Average score on the MFIS-5 fatigue impact measure, across participants
MFIS-5 Mean Score at 5 weeks | 5 weeks from date of consent
  Average score on the MFIS-5 fatigue impact measure, across participants
MFIS-5 Mean Score at 10 weeks | 10 weeks from date of consent
  Average score on the MFIS-5 fatigue impact measure, across participants
MFIS-5 Standard Deviation of Mean Score at 0 weeks | 0 weeks from date of consent
  Standard deviation around Mean Score on MFIS-5 fatigue impact measure across participants
MFIS-5 Standard Deviation of Mean Score at 5 weeks | 5 weeks from date of consent
  Standard deviation around Mean Score on MFIS-5 fatigue impact measure across participants
MFIS-5 Standard Deviation of Mean Score at 10 weeks | 10 weeks from date of consent
  Standard deviation around Mean Score on MFIS-5 fatigue impact measure across participants
Depression Digital Visual Analogue Scale (VAS) Completion Rate (denominator is number consenting) at 0 weeks | 0 weeks from date of consent
  Percentage of those who consent to take part that complete the single digital VAS regarding severity of depression
Depression Digital Visual Analogue Scale (VAS) Completion Rate (denominator is number consenting) at 5 weeks | 5 weeks from date of consent
  Percentage of those who consent to take part that complete the single digital VAS regarding severity of depression
Depression Digital Visual Analogue Scale (VAS) Completion Rate (denominator is number consenting) at 10 weeks | 10 weeks from date of consent
  Percentage of those who consent to take part that complete the single digital VAS regarding severity of depression
Depression Digital Visual Analogue Scale (VAS) Mean Score at 0 weeks | 0 weeks from date of consent
  Average score on the 100 point digital VAS across participants
Depression Digital Visual Analogue Scale (VAS) Mean Score at 5 weeks | 5 weeks from date of consent
  Average score on the 100 point digital VAS across participants
Depression Digital Visual Analogue Scale (VAS) Mean Score at 10 weeks | 10 weeks from date of consent
  Average score on the 100 point digital VAS across participants
Depression Digital VAS Standard Deviation of Mean Score at 0 weeks | 0 weeks from date of consent
  Standard deviation around Mean Score on depression VAS across participants
Depression Digital VAS Standard Deviation of Mean Score at 5 weeks | 5 weeks from date of consent
  Standard deviation around Mean Score on depression VAS across participants
Depression Digital VAS Standard Deviation of Mean Score at 10 weeks | 10 weeks from date of consent
  Standard deviation around Mean Score on depression VAS across participants
Anxiety Digital Visual Analogue Scale (VAS) Completion Rate (denominator is number consenting) at 0 weeks | 0 weeks from date of consent
  Percentage of those who consent to take part that complete the single digital VAS regarding severity of anxiety
Anxiety Digital Visual Analogue Scale (VAS) Completion Rate (denominator is number consenting) at 5 weeks | 5 weeks from date of consent
  Percentage of those who consent to take part that complete the single digital VAS regarding severity of anxiety
Anxiety Digital Visual Analogue Scale (VAS) Completion Rate (denominator is number consenting) at 10 weeks | 10 weeks from date of consent
  Percentage of those who consent to take part that complete the single digital VAS regarding severity of anxiety
Anxiety Digital VAS Mean Score at 0 weeks | 0 weeks from date of consent
  Average score on the 100 point digital VAS across participants
Anxiety Digital VAS Mean Score at 5 weeks | 5 weeks from date of consent
  Average score on the 100 point digital VAS across participants
Anxiety Digital VAS Mean Score at 10 weeks | 10 weeks from date of consent
  Average score on the 100 point digital VAS across participants
Anxiety Digital VAS Standard Deviation of Mean Score at 0 weeks | 0 weeks from date of consent
  Standard deviation around Mean Score on the Anxiety digital VAS across participants
Anxiety Digital VAS Standard Deviation of Mean Score at 5 weeks | 5 weeks from date of consent
  Standard deviation around Mean Score on the Anxiety digital VAS across participants
Anxiety Digital VAS Standard Deviation of Mean Score at 10 weeks | 10 weeks from date of consent
  Standard deviation around Mean Score on the Anxiety digital VAS across participants
Sleep Condition Index (SCI) Completion Rate (denominator is number consenting) at 0 weeks | 0 weeks from date of consent
  Percentage of those who consent to take part that complete all 8 questions of the SCI
Sleep Condition Index (SCI) Completion Rate (denominator is number consenting) at 5 weeks | 5 weeks from date of consent
  Percentage of those who consent to take part that complete all 8 questions of the SCI
Sleep Condition Index (SCI) Completion Rate (denominator is number consenting) at 10 weeks | 10 weeks from date of consent
  Percentage of those who consent to take part that complete all 8 questions of the SCI
Sleep Condition Index (SCI) Mean Score at 0 weeks | 0 weeks from date of consent
  Average score on the SCI across participants
Sleep Condition Index (SCI) Mean Score at 5 weeks | 5 weeks from date of consent
  Average score on the SCI across participants
Sleep Condition Index (SCI) Mean Score at 10 weeks | 10 weeks from date of consent
  Average score on the SCI across participants
Sleep Condition Index (SCI) Standard Deviation of Mean Score at 0 weeks | 0 weeks from date of consent
  Standard deviation around Mean Score on the SCI across participants
Sleep Condition Index (SCI) Standard Deviation of Mean Score at 5 weeks | 5 weeks from date of consent
  Standard deviation around Mean Score on the SCI across participants
Sleep Condition Index (SCI) Standard Deviation of Mean Score at 10 weeks | 10 weeks from date of consent
  Standard deviation around Mean Score on the SCI across participants
PAM-10 Completion Rate (denominator is number consenting) at 0 weeks | 0 weeks from date of consent
  Percentage of those who consent to take part that complete all 10 questions of the Patient Activation Measure (PAM-10)
PAM-10 Completion Rate (denominator is number consenting) at 5 weeks | 5 weeks from date of consent
  Percentage of those who consent to take part that complete all 10 questions of the Patient Activation Measure (PAM-10)
PAM-10 Completion Rate (denominator is number consenting) at 10 weeks | 10 weeks from date of consent
  Percentage of those who consent to take part that complete all 10 questions of the Patient Activation Measure (PAM-10)
PAM-10 Mean Score at 0 weeks | 0 weeks from date of consent
  Average score on the PAM-10 across participants
PAM-10 Mean Score at 5 weeks | 5 weeks from date of consent
  Average score on the PAM-10 across participants
PAM-10 Mean Score at 10 weeks | 10 weeks from date of consent
  Average score on the PAM-10 across participants
PAM-10 Standard Deviation of Mean Score at 0 weeks | 0 weeks from date of consent
  Standard deviation around Mean Score on the PAM-10 across participants
PAM-10 Standard Deviation of Mean Score at 5 weeks | 5 weeks from date of consent
  Standard deviation around Mean Score on the PAM-10 across participants
PAM-10 Standard Deviation of Mean Score at 10 weeks | 10 weeks from date of consent
  Standard deviation around Mean Score on the PAM-10 across participants
User Demographics | 0 weeks from date of consent
  Investigator-developed questionnaire asking users to enter their gender (M/F/Other/Prefer not to say), age (years), whether users have primary or secondary Sjogren's syndrome, number of years since diagnosis, country of residence, and any other conditions users wish to report.

SECONDARY OUTCOMES:
App user retention | Interaction data will be collected continuously for up to 13 weeks for each participant.
  Percentage of participants who launch the app at least once a week as recorded by automatically-generated logs
Frequency of app engagement | Interaction data will be collected continuously for up to 13 weeks for each participant.
  The maximum, minimum and average number of times the app is launched
Duration of app engagement | Interaction data will be collected continuously for up to 13 weeks for each participant.
  The maximum, minimum and average length of time users interact with app
Depth of app engagement | Interaction data will be collected continuously for up to 13 weeks for each participant.
  The maximum, minimum and average number of times users interact with specific app features after launching the app
Acceptability of app and study procedures | Interviews will take place after users have had the app installed on their device for 10 weeks after date of consent
  All users will be invited to participate in a remote qualitative interview (up to 60 minutes). We do not expect that all participants will take part, and aim to recruit n=20 (10 in experimental group, 10 in control group). Interested users will be contacted via email to consent and arrange a suitable interview time. Semi-structured interviews will explore acceptability of the app and study procedures (i.e. affective attitude, burden, perceived effectiveness of the app, ethicality, app coherence, and opportunity costs) and usability of the app (informed by items on the System Usability Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Katie L Hackett, PhD, Principal Investigator — Northumbria University; Claire H McCallum, PhD, Study Chair — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data sets (including answers to questionnaires, smartphone interaction data, and qualitative interview data) may be used to support future student projects at Northumbria University, however these datasets will be fully anonymised before being shared.